CLINICAL TRIAL: NCT05022160
Title: Preventing Catheter Related Bladder Discomfort (CRBD) in Male Patients Undergoing Lower Urinary Tract Surgery With Bilateral Pudendal Nerve Block: a Randomized Control Trial
Brief Title: Preventing Catheter Related Bladder Discomfort (CRBD) With Bilateral Pudendal Nerve Block
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Principal Investigator, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uro-Adm-Trg-1/IRB/2021/122
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Bladder Neoplasm; Prostatic Neoplasms
Keywords: Bupivacaine; pudendal nerve block; CRBD
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Experimental): Patients in this group will receive bilateral pudendal nerve block after spinal anesthesia- before starting the surgery
  Interventions: Drug: pudendal nerve block
- Group C (Placebo Comparator): Patients in this group will only receive spinal anesthesia before starting the surgery
  Interventions: Drug: pudendal nerve block

INTERVENTIONS:
Drug: pudendal nerve block — All patients in the study group will receive bilateral pudendal nerve block at the end of surgery, with help of landmark technique, using 0.5% bupivacaine

SUMMARY:
Bladder irrigation with a 3 way foley catheter is an important component of post operative management of transurethral bladder surgeries. But it is associated with a high incidence of bladder discomfort. Catheter related bladder discomfort (CRBD) doesn't respond to the orthodox opioid pain medication and is greatly distressful to the patients postoperatively, adversely affecting the quality of recovery often requiring administration of additional pain medication thereby increasing treatment costs, patient dissatisfaction and longer hospital stays. Several systemic agents have been used to reduce CRBD, but they have many side effects. A trial has been planned to find a way of reducing CRBD avoid distressing systemic side effects

DETAILED DESCRIPTION:
INTRODUCTION:

Trans urethral resection of prostate (TURP) and trans urethral resection of bladder tumor (TURBT) are the two most commonly performed endourological procedures associated with complication rates of 10% and 11% respectively.1 This relatively high percentage of complications can be owed to the amount of blood loss that occurs in these surgical procedures and can cause subsequent clot retention. Irrigation attached with three-way large bore urinary catheters is employed in order to avoid this clot retention.2 Catheter related bladder discomfort (CRBD) is a consequence of these large bore urinary catheters irritating the bladder mucosa causing involuntary bladder contractions being mediated by urothelial muscarinic receptors.3 The incidence of CRBD ranges from 47% to 90%.4 CRBD induced by indwelling urinary catheter is characterized by supra-pubic discomfort and a burning sensation in the urethra accompanied by an intense urge to void and increased urinary frequency.5 CRBD doesn't respond to the orthodox opioid pain medication and is greatly distressful to the patients postoperatively, adversely affecting the quality of recovery often requiring administration of additional pain medication thereby increasing treatment costs, patient dissatisfaction and longer hospital stays.3-5 The sensory supply of urethra and bladder neck is carried by Pudendal nerve. It originates from the ventral rami of the anterior nerve roots arising from sacral segments S2 to S4. Therefore theoretically, CRBD can be prevented by applying Pudendal Nerve Block (PNB).5 Xiaoqiang et al in 2017 reported that pudendal nerve block significantly reduced incidence of post-operative CRBD with administration of pudendal nerve block as compared to controls. The frequency of postoperative CRBD was at 63% in PNB versus 82% in control group at 30 minutes which was statistically significant (p=0.004). Similarly, the frequency of CRBD at 2 hours was 64% in PNB and 90% in control group (p˂0.001); and the frequency of CRBD at 8 hours was 58% in PNB and 79% in control group (p=0.003) respectively coinciding with the duration of action of Ropivacaine. Beyond that time there was no statistically significant difference between the two groups.5

RATIONALE:

The rationale of this study is that there is no previous study on this specific topic in the Pakistan. Thus, the findings of my study will help to determine the efficacy of pudendal nerve block in preventing CRBD in our population and will help improve evidence-based practices in patients undergoing TURP and TURBT.

OBJECTIVES:

"To compare between spinal anesthesia with pudendal nerve block versus spinal anesthesia alone in terms of frequency of post-operative CRBD and its severity in patients undergoing TURP and TURBT"

OPERATIONAL DEFINITIONS:

1. CATHETER RELATED BLADDER DISCOMFORT CRBD will be defined as presence of supra-pubic discomfort and a burning sensation in the urethra accompanied by an intense urge to void.
2. PUDENDAL NERVE BLOCK PNB is achieved by Infiltration of .5% ropivacaine in 5ml increments, maximum of 10 ml bilaterally, around Pudendal nerve on both sides under nerve stimulator guidance via two separate punctures 3 and 9 o'clock; approximately 3.5 to 4 cm from the center of the anus after making lithotomy position and aseptic preparation of the skin.
3. NUMERIC RATING SCALE FOR PAIN Numeric Rating Scale for Pain (NRSP) is a continuous scale of pain intensity, consisting of a straight line 10 cm long between the two end-points from 0-10. The patient will specify their level of pain by indicating a position along this line, as detailed in Annexure C. Pain will be scored as no pain (0), mild pain (<4 cm), moderate pain (4-7 cm) and severe pain (>7 cm).

HYPOTHESIS:

Spinal anesthesia and Pudendal Nerve Block are better than spinal anesthesia alone in preventing post-operative CRBD in patients undergoing TURP and TURBT.

MATERIAL AND METHODS:

1. STUDY DESIGN: Randomized controlled clinical trial.
2. SETTING: Armed Forces Institute of Urology, Rawalpindi.
3. DURATION OF STUDY: 6 Months after approval of synopsis
4. SAMPLE SIZE: Sample size calculated using WHO sample size calculator

   1. Power of Test = 95%.
   2. Level of Significance = 5%
   3. Anticipated population proportion 1 = 63% 5
   4. Anticipated population proportion 2 = 82% 5
   5. Minimum sample size in each group (n) = 125 patients in each group.
   6. Total Sample size = 250 patients.
5. SAMPLING TECHNIQUE: Non-probability consecutive sampling.

SAMPLE SELECTION:

1. INCLUSION CRITERIA:

   1. Male patients.
   2. Age >18 years
   3. Patients undergoing TURP & TURBT
   4. No history of chronic pain
   5. ASA I, II & III
2. EXCLUSION CRITERIA:

   1. Female gender
   2. Ischemic Heart Disease
   3. Chronic Obstructive Pulmonary Disease
   4. Coagulopathy
   5. Mental Disorder
   6. ASA IV & V The above-mentioned factors will act as confounders introducing bias in the study thus excluded.

DATA COLLECTION PROCEDURE:

A Total of 250 patients from Armed Forces Institute of Urology, Rawalpindi undergoing TURP or TURBT who will meet the inclusion and exclusion criterion will be enrolled in the study after taking permission from hospital ethical review committee and approval of synopsis from CPSP REU. Written informed consent will be taken from patients included in the study attached as Annexure A.

Patients will be randomly divided into 2 groups; group A and group B containing 125 patients each by lottery method. Group A patients will be administered bilateral pudendal nerve block with 0.5% Ropivacaine after giving spinal anesthesia while group B patients will only be given spinal anesthesia before undergoing TURP or TURBT.

Patient demographics will be documented before the surgery. Postoperatively all the patients will be observed at intervals of 30 minutes, 08 and 24 hours for development of any post-operative CRBD and its severity. Data in both the groups will be recorded on a predesigned proforma of questionnaire attached in the end as Annexure B.

All patients will be given due respect and their comfort will be taken care of during examination. The exclusion criteria will be strictly followed to control confounders and bias in the study.

DATA ANALYSIS PLAN:

Data will be entered in and analyzed by SPSS Version 16. Mean and standard deviation will be calculated for the quantitative variables i.e. Age, BMI etc. Qualitative variables like gender, ASA grade and CRBD severity will be expressed as frequency and percentages. Effect modifiers like age, BMI and ASA grade will be controlled by stratification. Frequency of CRBD in both the groups will be compared by applying post stratification Chi square test. P value ≤ 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Male patients.
* Age >18 years
* Patients undergoing TURP & TURBT under spinal anesthesia
* No history of chronic pain
* ASA I, II & III

Exclusion Criteria:

* Female gender
* Ischemic Heart Disease
* Chronic Obstructive Pulmonary Disease
* Coagulopathy
* Mental Disorder
* ASA IV & V
* Conversion of spinal anesthesia to general anesthesia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Catheter related bladder discomfort | 24 hours post surgery
  Frequency of catheter related bladder discomfort at 3,8,12 and 24 hours after surgery

SECONDARY OUTCOMES:
average intensity of Catheter related bladder discomfort | 24 hours post surgery
  average intensity of CRBD using numeric rating scale for pain at 3,8,12 and 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Madiha Ahmed, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel HD, Ball MW, Cohen JE, Kates M, Pierorazio PM, Allaf ME. Morbidity of urologic surgical procedures: an analysis of rates, risk factors, and outcomes. Urology. 2015 Mar;85(3):552-9. doi: 10.1016/j.urology.2014.11.034. PMID 25733265
- [Background] Xiaoqiang L, Xuerong Z, Juan L, Mathew BS, Xiaorong Y, Qin W, Lili L, Yingying Z, Jun L. Efficacy of pudendal nerve block for alleviation of catheter-related bladder discomfort in male patients undergoing lower urinary tract surgeries: A randomized, controlled, double-blind trial. Medicine (Baltimore). 2017 Dec;96(49):e8932. doi: 10.1097/MD.0000000000008932. PMID 29245259